CLINICAL TRIAL: NCT06453265
Title: A Double-Blind, Randomized, Crossover Study to Assess the Abuse Potential of Intranasal Cebranopadol Compared to Oxycodone and Placebo in Healthy, Nondependent Recreational Opioid Users
Brief Title: A Study to Assess the Abuse Potential of Intranasal Cebranopadol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRN-228-102
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Abuse, Drug
Keywords: Human Abuse Potential
MeSH Terms: conditions — Substance-Related Disorders | interventions — 6'-fluoro-4',9'-dihydro-N,N-dimethyl-4-phenylspiro(cyclohexane-1,1'(3'H)-pyrano(3,4-b)indol)-4-amine

STUDY DESIGN:
Intervention Model Description: Assessment of the Abuse Potential of Intranasal Cebranopadol Compared to Oxycodone and Placebo in Healthy, Nondependent Recreational Opioid Users
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Selection- 600ug (Part A) (Experimental): Cebranopadol 600 ug single dose
  Interventions: Drug: Cebranopadol- 600 ug
- Dose Selection - 800 ug (Part A) (Experimental): Cebraopadol 800 ug single dose
  Interventions: Drug: Cebranopadol- 800ug
- Dose Selection- 1000 ug (Part A) (Experimental): Cebranopadol 1000 ug single dose
  Interventions: Drug: Cebranopadol- 1000ug
- Qualification Phase - Oxycodone (Part B) (Active Comparator): Oxycodone 40mg
  Interventions: Drug: Qualification
- Qualification Phase - Placebo (Part B) (Placebo Comparator): Matching Placebo
  Interventions: Drug: Qualification
- Treatment Phase A- (Part B) (Experimental): -Treatment A: Cebranopadol
  Interventions: Drug: Treatment A:
- Treatment Phase B- (Part B) (Active Comparator): - Treatment B: Oxycodone HCl IR 40 mg
  Interventions: Drug: Treatment B
- Treatment Phase C (Part B) (Placebo Comparator): - Treatment C: Placebo
  Interventions: Drug: Treatment C

INTERVENTIONS:
Drug: Cebranopadol- 600 ug — Dose ascending cohorts
  - Cebranopadol 600 ug single dose
  Arms: Dose Selection- 600ug (Part A)
Drug: Cebranopadol- 800ug — Dose ascending cohorts
  - Cebraopadol 800 ug single dose
  Arms: Dose Selection - 800 ug (Part A)
Drug: Cebranopadol- 1000ug — Dose ascending cohorts
  - Cebranopadol 1000 ug single dose
  Arms: Dose Selection- 1000 ug (Part A)
Drug: Treatment A: — Cebranopadol, dose determined in Part A
  Arms: Treatment Phase A- (Part B)
Drug: Treatment B — Oxycodone HCl IR 40 mg
  Arms: Treatment Phase B- (Part B)
Drug: Treatment C — Placebo
  Arms: Treatment Phase C (Part B)
Drug: Qualification — Oxycodone 40mg
  Arms: Qualification Phase - Oxycodone (Part B)
Drug: Qualification — Matching Placebo
  Arms: Qualification Phase - Placebo (Part B)

SUMMARY:
The purpose of this study to Assess the Abuse Potential of Intranasal Cebranopadol Compared to Oxycodone and Placebo in Healthy, Nondependent Recreational Opioid Users.

DETAILED DESCRIPTION:
This study will be conducted to examine the intranasal abuse potential of cebranopadol compared with oxycodone HCl IR and placebo in recreational opioid users with intranasal experience, a Dose Escalation Phase (Part A) will first be conducted to determine a safe dose for evaluation in the Main Study (Part B).

The Dose Selection Phase (Part A) will consist of 3 phases: Screening, Treatment and Follow-up. Subjects will participate in an outpatient medical screening visit, a 4-day treatment visit and a follow-up phone call.

The Main Study (Part B) will consist of 4 phases: Screening, Qualification, Treatment and Follow-up. Subjects will participate in an outpatient screening visit, a 4-day Qualification Phase, a 30-day Treatment Phase and a follow-up phone call.

ELIGIBILITY:
Key Inclusion Criteria:

* Experienced opioid user who meets the following criteria: (1) has used opioids for nontherapeutic purposes (i.e., for psychoactive effects) on at least 10 occasions in the year prior to Screening; (2) has used opioids at least once in the 12 weeks prior to Screening; and (3) self-reported intranasal use of drugs of abuse on at least 3 occasions in the year prior to Screening.
* Subjects must be in good health as determined by medical history, physical examination, 12-lead ECG and vital signs measures (pulse rate, systolic and diastolic blood pressure, respiratory rate and oxygen saturation using pulse oximetry) at Screening.
* Subjects must be willing to comply with the requirements and restrictions of the study.

Key Exclusion Criteria:

* Drug or alcohol dependence in the 12 months prior to Screening (except nicotine), as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR), or any self-reported dependence or "addiction" within the subject's lifetime (except nicotine or caffeine).
* Subjects who have ever been in treatment for substance use disorder(s) (except smoking cessation).
* History or presence of any clinically significant cardiac, psychiatric, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, renal or other disease at Screening, which, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results.
* Clinically significant abnormalities in the intranasal cavity (including a deviated septum, perforated nasal septum, rhinorrhea, or excessive sneezing) or any condition that, in the opinion of the investigator, would interfere with the study procedures, data integrity or would compromise the safety of the subject. Subjects with nasal piercings/nose rings will be required to remove them for the duration of their inpatient stay.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Drug Liking VAS Emax | 48 hrs of Tmax for each treatment
  The primary pharmacodynamic endpoint (Drug Liking VAS Emax) will be evaluated with a linear mixed-effects model, containing treatment, period, sequence and first-order carryover as fixed effects and subject nested within sequence as random effect, using the Modified Completer Population

CONTACTS AND LOCATIONS:
Overall Officials: Angela Eakin, MD, Principal Investigator — Ohio Clinical Trials
Locations (1):
- Ohio Clinical Trials, Inc., Columbus, Ohio, United States